CLINICAL TRIAL: NCT00000303
Title: Rapid Evaluation of Cocaine Pharmacotherapies (Baclofen)
Brief Title: Rapid Evaluation of Baclofen for Treatment of Cocaine Abuse/Dependence - 6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09260-6; P50DA009260 (NIH); P50-09260-6
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Baclofen

INTERVENTIONS:
Drug: Baclofen

SUMMARY:
The purpose of this study is to empirically test a series of medications to: 1) determine each medication's efficacy in treatment of cocaine abuse/dependence; 2) find most effective dose range for each medication. In this study, baclofen is tested.

DETAILED DESCRIPTION:
16-week participation plus a 2 week lead in period. Participants are assigned randomly to placebo or baclofen. Participant attend group meetings 3 x/week.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 18-65. cocaine dependence according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria. Self-reported use within the last 30 days. Agreeable to conditions of study and signed informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy, history of seizures, pregnant and/or nursing women, dependence on ethanol (ETOH) or benzodiazepines or other sedative-hypnotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1997-10; Primary Completion 1999-05 (Actual)

PRIMARY OUTCOMES:
Retention
Cocaine use
Cocaine craving
Psychosocial progress

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States